CLINICAL TRIAL: NCT03076346
Title: Neural Biomarkers of Clozapine Response
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Deepak K. Sarpal, M.D., MD, University of Pittsburgh
Other Study IDs: STUDY19060115
Record Dates: First submitted 2017-03-06; First posted 2017-03-10 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Schizophrenia; Treatment-resistant Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Schizophrenia, Treatment-Resistant; Psychotic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Clozapine has consistently shown to be a superior drug for psychosis in patients who do not respond to other treatments, but its mechanism of action remains unknown. The overall goal of this study is to examine the functional neural circuitry that underlies successful treatment with clozapine, which may lead to the identification of biomarkers that will allow for more efficient use of clozapine, as well as additional treatment targets for patients with refractory illness.

DETAILED DESCRIPTION:
A large number of patients with chronic psychotic disorders continue to have symptoms following unsuccessful trials with first-line antipsychotic drugs. For these patients with refractory psychosis, clozapine has consistently demonstrated superior efficacy. Clozapine is often underutilized and administered late in a patient's course of treatment, which leads to increased morbidity, unnecessary medication trials, and increased health care expenditure. Meanwhile, the mechanism of action underlying clozapine's novel effects remains unknown and has not been studied with modern neuroimaging methods. Identifying the neural mechanisms by which clozapine exerts its effects may lead to biomarkers that will facilitate efficient utilization of the drug, and introduce novel treatment targets. In patients with refractory psychotic symptoms, the proposed study will use resting-state and task-based functional MRI (fMRI) to examine the neural circuitry of efficacious treatment with a trial of clozapine. Patients will undergo fMRI scanning both before and after 12 weeks of treatment, with the aims of determining: baseline patterns of resting-state functional connectivity and task-based activation that predict response to treatment; and changes in resting-state and task-based functional circuitry associated with efficacious treatment. Results of this proposal may lead to biomarkers that will optimize treatment algorithms for psychotic disorders and facilitate drug development for refractory psychosis.

ELIGIBILITY:
Inclusion Criteria:

1. Current positive symptoms rated ≥4 (moderate) on one or more of these Brief Psychiatric Rating Scale items: hallucinatory behavior, unusual thought content and conceptual disorganization.
2. Patient has failed two trials of treatment with antipsychotic drugs and the patient's clinical team is initiating clozapine.
3. Age of 18 to 50.
4. Patient is competent and willing to sign informed consent.
5. For female patients, negative pregnancy test and agreement to use a medically accepted birth control method.
6. Diagnosis of schizophrenia or schizoaffective disorder

Exclusion Criteria:

1. Serious neurological or endocrine disorder.
2. Any medical condition which requires treatment with a medication with psychotropic effects
3. Significant risk of suicidal or homicidal behavior
4. Cognitive or language limitations, or any other factor that would preclude subjects providing informed consent
5. Contraindications to treatment with clozapine (e.g. failed response in past, or history of adverse reactions to treatment).
6. Contraindications to magnetic resonance imaging (e.g. pacemaker).
7. Female patients who are pregnant or breast feeding.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with schizophrenia or schizoaffective disorder who have failed treatment with two antipsychotic drugs and are beginning treatment with clozapine.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in resting state functional connectivity with efficacious clozapine treatment | 12 weeks
  The investigators will examine the functional circuitry associated with a reduction of psychotic symptoms assessed with the Brief Psychiatric Rating Scale.

SECONDARY OUTCOMES:
Baseline prediction of clozapine response | 12 weeks
  The investigators will use a pattern of baseline functional connectivity to predict successful reduction of psychotic symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Wpic/Upmc, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No